CLINICAL TRIAL: NCT04811950
Title: Assessment of Prognostic Role of Platelet-lymphocyte and Neutrophil _monocyte Ratio in CLL
Brief Title: Prognostic Role of Platelet _lymphocyte and Neutrophil _monocyte in CLL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Hussein Mahmoud, Principal investigator, Assiut University
Other Study IDs: Prognostic factors in CLL
Record Dates: First submitted 2019-09-30; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: CLL Progression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Emerald — Complete blood countdevice

SUMMARY:
The biological rationale in calculating PLR stems from the increase in the lymphocyte count and reduction in the platelet count often encountered in the advances stages of CLL .NMR median value was significantly higher in untreated patients than in patients who received treatment strengthening the hypothesis that this ratio is associated with a more indolent form of disease

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common type of leukemia in the western world. In Egypt, CLL is the most common subtype of leukemias

* the National Cancer Registry reported over 80% of lymphoid leukemias are CLL . It is the most common types of leukemia diagnosed in adult. ChroniclymphocyticleukemialymphocytesareclonalCD19-positiveBcells characterized by the accumulation of CD5 positive monoclonal B cells in peripheral blood. Bone marrow aspiration shows lymphocytic replacement of normal marrow elements, lymphocytes comprise 25-95% .Trephine biopsy reveals nodular, diffuse or interstitial involvement by lymphocytes
* Both the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) and European Society of Medical Oncology guidelines also require persistence of lymphocytosis for longer than 3 months

The most important prognostic factors in CLL are clinical staging systems developed by Rai and Binet

. These systems based on clinical examination e.g. lymphadenopathy and organomegaly, peripheral blood findings (platelet andhaemoglobinvalues),markersoftumorload(thymidinekinaseand B2-microglobulin), expression of specific proteins in CLL cells; CD38, CD49d & ZAP-70, genetic abnormalities quantified by FISH which include del(13q), tri12, del(11q), & del(17p) and genetic parameters.including immunoglobulin heavy chain variable gene segment (IGHV) mutational status. Finally, prognostication in patients with CLL should not only address disease progression and overall survival, but also response to therapy. The biological rationale in calculating PLR stems from the increase in the lymphocyte count and reduction in the platelet count often encountered in the advanced stages of CLL. Therefore, we hypothesized that the ratio using both the platelet and lymphocyte counts may have a prognostic role in patients with CLL. Neutrophil-monocyte ratio(NMR) was found to be higher in untreated patients than in patients who received treatment . and therefore it will be used to prove its relation with disease severity and itsprognosticvalues. It is important to highlight that using these indices, is simple, cheap, easily measured and reproducible and can be integrated into our daily clinical practice as prognostic marker of CLL

ELIGIBILITY:
Inclusion Criteria:

- All CLL patients

Exclusion Criteria:

* CLL patients on treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients with CLL come to South Egypt Cancer institute from 2010 to 2020
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
platelet-lymphocyte and neutrophilo_monocyte ratio in CLL | base line
  Calculating the ratio of platelets to lymphocytes and neutrophils to monocytes in CLL cases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu H, Xu W, Shen QD. [Serum levels of soluble CD(23) and thrombopoietin in chronic lymphocytic leukemia]. Zhonghua Nei Ke Za Zhi. 2008 Oct;47(10):826-9. Chinese. PMID 19080142